CLINICAL TRIAL: NCT00075088
Title: Tele-electrocardiography in Emergency Cardiac Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1R01NR007881-01A2 (NIH); R01NR007881 (NIH); NCT00305318 (obsolete NCT alias)
Record Dates: First submitted 2004-01-02; First posted 2004-01-05 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-05

CONDITIONS: Myocardial Infarction; Chest Pain
Keywords: Telemedicine; Emergency Care; Cardiac
MeSH Terms: conditions — Myocardial Infarction; Chest Pain | interventions — Electrocardiography; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrocardiogram (ECG) Intervention (Experimental): Patients randomized to the experimental group had their ECGs printed out in the target ED with an audible voice alarm. Print-out of the pre-hospital ECG in the target ED was the intervention.
  Interventions: Device: Electrocardiogram (ECG) Intervention
- Routine Clinical Practice (Other): Control patients had an ECG conducted after hospital arrival, as was the standard of care in the county.
  Interventions: Other: Routine Clinical Practice

INTERVENTIONS:
Device: Electrocardiogram (ECG) Intervention — Pre-hospital electrocardiographic (ECG) monitoring with special software to detect myocardial ischemia and to automatically transmit an ECG to the destination hospital emergency department with a voice alarm announcing "Incoming ECG from the field" and print out in the ED.
  Arms: Electrocardiogram (ECG) Intervention
Other: Routine Clinical Practice — ECG in the ED as part of routine clinical practice.
  Arms: Routine Clinical Practice

SUMMARY:
The purpose of this study is to see whether individuals who access the "911" emergency medical system with a heart attack or severe chest pain will receive more timely hospital treatment and better outcomes if hospital clinicians are provided with earlier and more complete electrocardiography (ECG) information.

DETAILED DESCRIPTION:
This is a Phase III study. Patients will be randomized (like tossing a coin) to 1 of 2 groups: Group 1: Patients will have pre-hospital ECG intervention. Group 2: Patients will have routine emergency heart care. Information will be collected about time symptoms started, clinical management, and other measures. All patients will be contacted by telephone 12 months later and interviewed as to whether they experienced any cardiac symptoms.

ELIGIBILITY:
Inclusion Criteria:

* All individuals in Santa Cruz County in California who call 911 with symptoms of acute coronary syndrome (chest pain, shortness of breath, anginal equivalent).

Exclusion Criteria:

* Those who don't meet the above inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 794 (Actual)
Dates: Start 2003-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Drew, RN PhD FAAN, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Drew BJ, Sommargren CE, Schindler DM, Benedict K, Zegre-Hemsey J, Glancy JP. A simple strategy improves prehospital electrocardiogram utilization and hospital treatment for patients with acute coronary syndrome (from the ST SMART Study). Am J Cardiol. 2011 Feb 1;107(3):347-52. doi: 10.1016/j.amjcard.2010.09.027. PMID 21256997
- [Result] Zegre Hemsey JK, Dracup K, Fleischmann K, Sommargren CE, Drew BJ. Prehospital 12-lead ST-segment monitoring improves the early diagnosis of acute coronary syndrome. J Electrocardiol. 2012 May-Jun;45(3):266-71. doi: 10.1016/j.jelectrocard.2011.10.004. Epub 2011 Nov 23. PMID 22115367
- [Result] Zegre-Hemsey J, Sommargren CE, Drew BJ. Initial ECG acquisition within 10 minutes of arrival at the emergency department in persons with chest pain: time and gender differences. J Emerg Nurs. 2011 Jan;37(1):109-12. doi: 10.1016/j.jen.2009.11.004. Epub 2009 Dec 11. PMID 21237383
- [Result] Drew BJ, Dempsey ED, Joo TH, Sommargren CE, Glancy JP, Benedict K, Krucoff MW. Pre-hospital synthesized 12-lead ECG ischemia monitoring with trans-telephonic transmission in acute coronary syndromes: pilot study results of the ST SMART trial. J Electrocardiol. 2004;37 Suppl:214-21. doi: 10.1016/j.jelectrocard.2004.08.060. PMID 15534844
- [Result] Drew BJ, Sommargren CE, Schindler DM, Zegre J, Benedict K, Krucoff MW. Novel electrocardiogram configurations and transmission procedures in the prehospital setting: effect on ischemia and arrhythmia determination. J Electrocardiol. 2006 Oct;39(4 Suppl):S157-60. doi: 10.1016/j.jelectrocard.2006.05.033. PMID 17015064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For 5-years, paramedics responding to 911 calls for symptoms suggestive of Acute Coronary Syndrome (ACS) in one U.S. county transmitted an electrocardiogram (ECG) to the target emergency department (ED) for all patients meeting eligibility criteria. A central computer received the transmission and randomized to an experimental or control group.
Pre-assignment Details: 4,219 calls to 911 for ACS symptoms were made over the study period; 3,103 pre-hospital ECGs were transmitted by paramedics; 2,353 ECGs were successfully received by the target emergency department (ED); 794 patients consented. If patient consent was not obtained, data were not used.
Period: Overall Study
Arm/Group | Electrocardiogram (ECG) Intervention | Routine Clinical Practice
Started | 403 | 391
Completed | 403 | 391
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electrocardiogram (ECG) Intervention | Routine Clinical Practice | Total
Number analyzed (Participants) | 403 | 391 | 794
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (15) | 71 (14) | 70 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 193 | 382
  Male | 214 | 198 | 412
Region of Enrollment [Number; unit: participants]
  United States | 403 | 391 | 794

OUTCOME MEASURES:

1. Primary Outcome: Hospital Time to Treatment for Patients With Unstable Angina/Non-STEMI
Description: Time from ED arrival to first drug was determined as recommended by American College of Cardiology/American Heart Association 2007 guidelines for management of patients with unstable angina/non-STEMI
Time Frame: Day 1
Population: Patients with unstable angina/non-STEMI. Four patients with Do Not Resuscitate (DNR) orders were excluded from this time-to-treatment analysis
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Electrocardiogram (ECG) Intervention | Routine Clinical Practice
Number analyzed (Participants) | 23 | 23
minutes | 23 (12) | 31 (16)

2. Primary Outcome: Hospital Time to Treatment for Patients With ST-elevation Myocardial Infarction (STEMI)
Description: Mean door-to-balloon time
Time Frame: Day 1
Population: 42 patients with STEMI who received primary percutaneous coronary intervention
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Electrocardiogram (ECG) Intervention | Routine Clinical Practice
Number analyzed (Participants) | 28 | 14
minutes | 78 (22) | 101 (56)

3. Secondary Outcome: Rehospitalization and Mortality
Time Frame: 4 years
Population: we did not have the resources to achieve this secondary aim that required long-term follow up (a labor intensive job). The PI is now retired.
Arm/Group | Electrocardiogram (ECG) Intervention | Routine Clinical Practice
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: Due to the low-risk intervention relative to participants' serious health condition, AEs were not collected if they did not meet the criteria for SAEs or were at least possibly attributable to study procedures (none were).
  Consented patients who died during the index hospitalization were reported. 786 were discharged alive.
Groups:
- Prehospital: At the start of the trial, the IRB requested every death in the pre-hospital period be reported because we put on the study electrocardiogram device in the field with waiver of consent so as not to cause a delay for patients reaching the hospital with possible heart attack. They were consented after they reached the hospital. However, IRB removed this requirement after 40 pre-consent/pre-hospital deaths were reported. The number of pre-hospital participants assessed before and after the IRB changed the reporting requirements cannot be determined from study data, but "NA" is not a valid entry in the "At Risk" field.
Arm/Group | Electrocardiogram (ECG) Intervention | Routine Clinical Practice | Prehospital
Serious Adverse Events (participants affected / at risk) | 5/403 | 3/391 | 40/40
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electrocardiogram (ECG) Intervention (N=403) | Routine Clinical Practice (N=391) | Prehospital (N=40)
Death (General disorders) | 5 (5) | 3 (3) | 40 (40)

LIMITATIONS AND CAVEATS:
Sample size was not powered to detect a statistically significant difference in survival between patients with and without a prehospital ECG

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes